CLINICAL TRIAL: NCT03774862
Title: Clinicopathological Importance of Colorectal Medullary Carcinoma: Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Serkan Zenger MD, General surgery specialist, V.K.V. American Hospital, Istanbul
Other Study IDs: VKVAmericanH
Record Dates: First submitted 2018-09-05; First posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Colorectal Medullary Carcinoma
Keywords: Medullary carcinoma; Colorectal cancer; Microsatellite instability
MeSH Terms: conditions — Carcinoma, Medullary; Colorectal Neoplasms; Microsatellite Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medullary carcinoma of colorectal cancers
- non-medullary carcinomas of the colorectal cancers

SUMMARY:
Medullary carcinoma (MC) is a rare tumor with solid growth pattern without glandular differentiation and constitute less than 1% of colorectal cancer. Lymph node positivity and distant organ metastasis were reported to be lower than other poorly differentiated adenocarcinomas. Therefore, the diagnosis of MC is pathologically important in terms of follow-up and treatment. MC is commonly localized in the right colon, has a large tumor size, and is mostly diagnosed in the T4 stage. As MC most likely have defects in DNA MMR, the correct pathological diagnosis is important for the postoperative treatment and the prognosis of the patients.

DETAILED DESCRIPTION:
427 patients with colorectal cancer who were underwent surgery between January 2011 and December 2017, were evaluated retrospectively into 2 groups as MC (n:13) and non-MC (n:414) in terms of demographic characteristics, pathological data and oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer diagnosis, medullary carcinoma

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 427 patients with colorectal cancer who were underwent surgery between January 2011 and December 2017, were evaluated retrospectively into 2 groups as MC (n:13) and non-MC (n:414) in terms of demographic characteristics, pathological data and oncological outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Overall survival of medullar colorectal carcinomas | 7 years

IPD SHARING:
Plan to Share IPD: No